CLINICAL TRIAL: NCT03767127
Title: Red Blood Cell Transfusion Decision Based on Arterial-venous Oxygen Difference Can Reduce Mortality in Critically Ill Patients
Brief Title: Oxygen Extraction-guided Transfusion in Critically Ill Patients
Status: Completed | Type: Observational
Sponsor: Università degli Studi di Ferrara (Other)
Responsible Party: Principal Investigator, Alberto Fogagnolo, Principal investigator, Università degli Studi di Ferrara
Other Study IDs: OEDT
Record Dates: First submitted 2018-11-30; First posted 2018-12-06 (Actual); Last update posted 2019-11-21 (Actual); Status verified 2019-11

CONDITIONS: Anemia; Critical Illness
Keywords: transfusion; intensive care medicine; 90-day mortality
MeSH Terms: conditions — Anemia; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Appropriate transfusion policy: Patients transfused with high arterial-venous oxygen difference (≥3.7 ml/dl) or non-transfused with low arterial-venous oxygen difference (<3.7 ml/dl)
- Non-Appropriate transfusion policy: Patients transfused despite low arterial-venous oxygen difference or non-transfused with high arterial-venous oxygen difference

SUMMARY:
Anemia is common in intensive care unit (ICU) patients and often appears early in the ICU course. The optimal management red blood cells RBC transfusion in critically ill patients remains controversial and clinical studies in this field have usually been based on transfusion thresholds. In the "TRICC" Trial, patients assigned to a restrictive transfusion strategy (transfusion if Hb<7 g/dL) had similar mortality to patients transfused if Hb<10 g/dL. Notably, none of the large RCT tried to focus on a personalize RBC transfusion protocol, i.e. a transfusion protocol which address the individual need for transfusion basing on physiological approach. We therefore hypothesized that patients with high extraction of oxygen could benefit more of RBCs transfusion regardless their hemoglobin levels.

ELIGIBILITY:
Inclusion Criteria:

* Hemoglobin level <10 g/dL during the first 72 hours of ICU

Exclusion Criteria:

* Acute bleeding
* Hemoglobin level less than 7 g/dL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Unselected critically ill patients admitted to intensive care unit
Sampling Method: Probability Sample
Enrollment: 177 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
90-day mortality | after 90 days from study enrollment
  mortality

SECONDARY OUTCOMES:
Acute kidney injury | 7 days after study inclusion
  Occurence of acute kidney injury according to KDIGO 2012 guidelines
Length of ICU stay | from ICU admission to discharge, up to 8 weeks
Variation in Sequential Organ Failure Assessment (SOFA) score | 5 days
  daily variation in SOFA score (0-24 points scale with higher values indicating worst conditions)
Days of vasopressor | 28 days after study inclusion
  Need for vasopressor

CONTACTS AND LOCATIONS:
Locations (1):
- Università di Ferrara, Ferrara, Italy

REFERENCES:
- [Derived] Fogagnolo A, Taccone FS, Vincent JL, Benetto G, Cavalcante E, Marangoni E, Ragazzi R, Creteur J, Volta CA, Spadaro S. Using arterial-venous oxygen difference to guide red blood cell transfusion strategy. Crit Care. 2020 Apr 20;24(1):160. doi: 10.1186/s13054-020-2827-5. PMID 32312299